CLINICAL TRIAL: NCT05085470
Title: Safety and Protective Efficacy of Repeated Controlled Human Schistosoma Mansoni Infection
Brief Title: Repeated Controlled Human Schistosoma Mansoni Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ReCoHSI
Record Dates: First submitted 2021-08-06; First posted 2021-10-20 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Schistosomiasis; Schistosoma Mansoni
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinfection group (Experimental): Participants will be exposed three times to 20 male Schistosoma mansoni cercariae (weeks 0, 9, and 18)
  Interventions: Biological: Schistosoma mansoni infection
- Infection control group (Active Comparator): 12 participants who will undergo a placebo mock infection with water twice (weeks 0 and 9) and will be exposed once to 20 male Schistosoma mansoni cercariae (week 18)
  Interventions: Biological: Schistosoma mansoni infection; Biological: Placebo mock infection

INTERVENTIONS:
Biological: Schistosoma mansoni infection — 20 viable male Schistosoma mansoni cercariae of the Puerto Rican strain
Biological: Placebo mock infection — Placebo mock infection with water
  Arms: Infection control group

SUMMARY:
A group of 24 healthy volunteers are challenged one or three times with 20 male Schistosoma mansoni cercariae to investigate whether this leads to protection and to identify potential correlates of protection

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits.
4. Subject will remain within Europe (excluding Corsica) during the study period.
5. Subject agrees to refrain from blood and plasma donation to Sanquin or for other purposes throughout the study period.
6. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
7. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, (severe) psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * body weight <50 kg or Body Mass Index (BMI) <18.0 or >35.0 kg/m2 at screening;
   * positive HIV, hepatitis B virus or hepatitis C virus screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
2. The chronic use of any drug known to interact with praziquantel, artesunate or lumefantrine metabolism (e.g. phenytoin, carbamazepine, phenobarbital, primidone, dexamethasone, rifampicin, cimetidine, flecainide, metoprolol, imipramine, amitriptyline, clomipramine, class IA and III anti-arrythmics, antipsychotics, antidepressants, macrolides, fluoroquinolones, imidazole- and triazole antimycotics, antihistamines). Because lumefantrine may cause extension of QT-time, chronic use of drugs with effect on QT interval will result in exclusion from study participation.
3. For female subjects: positive urine pregnancy test at screening.
4. Any history of schistosomiasis or treatment for schistosomiasis.
5. Positive serology for schistosomiasis or elevated serum CAA at screening.
6. Known hypersensitivity to or contra-indications (including co-medication) for use of praziquantel, artesunate or lumefantrine.
7. Being an employee or student of the department of Parasitology or Infectious diseases of the LUMC.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Protective efficacy | From week 18 until week 30
  The protective efficacy of repeated exposure to male Sm cercariae measured by the difference in frequency of serum circulating aniodic antigen (CAA) positivity (≥1.0 pg/mL) between the reinfection group and the infection control group at any timepoint after the final infection at week 18 and before week 30
Safety of (repeated) exposure to male Sm cercariae based on self-reported adverse events | 38 weeks
  Frequency and severity of adverse events after (repeated) human Sm infection with male cercariae

SECONDARY OUTCOMES:
Time to CAA positivity | From week 18 until week 30
  Comparison of time to positive serum and urine CAA test between the reinfection and infection control groups after the final infection at week 18 and before week 30
Peak serum CAA levels | From week 18 until week 30
  Comparison of peak serum CAA concentration between the reinfection and infection control group after the final infection at week 18 and before week 30
Eosinophils | From week 18 until week 30
  Comparison of eosinophil counts between the reinfection and infection control groups after challenge after the final infection at week 18 and before week 30
Antibody responses | From week 18 until week 30
  Comparison of (glycan) antibody responses directed against Sm antigens between the reinfection and infection control participants as well as between protected and non-protected participants after the final infection at week 18 and before week 30 using protein and glycan arrays
Cellular responses | From week 18 until week 30
  Comparison of cellular responses directed against Sm antigens between the reinfection and infection control participants as well as between protected and non-protected participants after the final infection at week 18 and before week 30 using flow cytometry
Attack rate | 26 weeks
  The pooled attack rate after initial exposure to 20 male cercariae, i.e. proportion CAA positivity between week 0-8 for the reinfection participants and between week 18-26 for infection control participants

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koopman JPR, Houlder EL, Janse JJ, Lamers OA, Roozen GV, Sijtsma JC, Casacuberta-Partal M, Hilt ST, van der Stoep MYEC, van Amerongen-Westra IM, Brienen EA, Wammes LJ, van Lieshout L, van Dam GJ, Corstjens PL, van Diepen A, Yazdanbakhsh M, Hokke CH, Roestenberg M. Clinical tolerance but no protective efficacy in a placebo-controlled trial of repeated controlled schistosome infection. J Clin Invest. 2024 Dec 12;135(4):e185422. doi: 10.1172/JCI185422. PMID 39666392